CLINICAL TRIAL: NCT02914171
Title: Phase I Safety and Feasibility Study of Intramyocardial Delivery of Autologous Bone Marrow Derived Mononuclear Cells to Right Ventricle of Patients With Ebstein Anomaly During Cardiac Surgery
Brief Title: Study of Autologous Bone Marrow Derived Mononuclear Cells for Treatment of Ebstein Anomaly
Acronym: Ebstein
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Timothy J. Nelson (Other)
Responsible Party: Sponsor-Investigator, Timothy J. Nelson, Program Director, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-007580
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Ebstein Anomaly
Keywords: Myopathic right ventricle
MeSH Terms: conditions — Ebstein Anomaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment arm (Experimental): Individuals with Ebstein anomaly and underlying myopathic right ventricle undergoing planned surgical intervention using an add-on procedure delivering autologous bone marrow-derived mononuclear cells into the right ventricle.
  Interventions: Biological: Autologous Bone Marrow-derived Mononuclear Cells; Device: Insertable cardiac monitor
- Control arm (Other): Individuals with Ebstein anomaly and underlying myopathic right ventricle undergoing planned surgical intervention without cell delivery.
  Interventions: Device: Insertable cardiac monitor

INTERVENTIONS:
Biological: Autologous Bone Marrow-derived Mononuclear Cells
  Other Names: MNC
  Arms: Treatment arm
Device: Insertable cardiac monitor — Following surgical Ebstein repair a Medtronic Reveal LINQ Insertable Cardiac Monitor (ICM) will be placed subcutaneously in the anterior chest to continuously monitor the subject's heart rhythm and to record cardiac information through automatic detection of arrhythmias.
  Other Names: ICM; ILR

SUMMARY:
The objective of this study is to determine the safety and feasibility of autologous mononuclear cells (MNS) collected from bone marrow (BM) and using an add-on intramyocardial delivery for individuals with Ebstein anomaly undergoing surgical intervention compared to the control group undergoing the same surgical procedure without cell delivery. This add-on procedure has the potential to foster a new strategy for individuals with congenital heart disease.This is an open-label study of autologous MNC derived from bone marrow with a 2-year follow-up to document 1) incidence and severity of adverse event and 2) monitor changes in cardiac structure and function.

DETAILED DESCRIPTION:
This study is an open label Phase I trial to determine the safety and feasibility of bone marrow-derived mononuclear cells to the right ventricle of subjects with Ebstein anomaly at the time of a planned surgical Ebstein repair compared to the control group undergoing the same planned surgical intervention without the cell delivery add-on procedure. Subjects will be screened at outpatient clinic visits at Mayo Clinic and interested qualified subjects will be consented and offered participation in this trial. Subject/Family will decide to participate in cell delivery or control arm. Once informed consent has been obtained, subjects will undergo identical evaluation (other than Hematology consultation and BM harvest occurring only in the cell-treatment group),preoperative values will be established/confirmed and a selection committee will review subjects within three days prior to planned procedure to confirm inclusion and exclusion criteria.However, individuals at high-risk, primarily neonates and those with preoperative advanced right heart failure will NOT be included such that the risk of this add-on procedure may not be acceptable. Following surgical Ebstein repair for the control group and following cell-based product delivery for the treatment group, all subjects will be followed for 24-months according to a pre-determined schedule that includes imaging studies along with a questionnaire, electrophysiology and laboratory studies at 1, 6, and 24 months post procedure. All subjects will be contacted for surveillance by phone at 3, 12, and 18 month post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 30 years
* Individuals clinically planned for elective surgical Ebstein repair
* Individuals able to undergo bone marrow aspirate according to clinical consultation with Hematology (cell treatment group only)
* Individuals able to undergo preoperative MRI or CT examination
* Individual and/or parent willing and able to give informed consent and willing to commit to completion of follow-up

Exclusion Criteria:

* Individuals requiring cavopulmonary shunt at the time of surgical Ebstein repair; planned preoperatively or required intraoperatively
* Individuals with, or reasonably expected to have, complications during surgical Ebstein repair or during post-operative recovery
* Individual who have not completed or will not be completing all pre-procedure work-up within 30 days of surgical Ebstein repair AND lack of pre-procedure work-up documented as a safety concern by a site investigator
* Individuals who have other clinical concerns as documented by a site investigator that could reasonably increase the risk of complications during or after surgical Ebstein repair
* Individuals whose cells have been determined, by the sponsor, to not be acceptable for release to the investigational site or individual whose cells have been compromised after cells released to investigational site (cell treatment group only)
* Individuals who require surgery on pulmonary, mitral, or aortic valve
* Individuals with pulmonary atresia or atrioventricular discordance with ventriculoarterial discordance
* Individuals with history of ventricular arrhythmia or new onset ventricular arrhythmia after enrollment that requires medical management
* Individuals who have undergone previous sternotomy
* Individuals with preoperative ventricular arrhythmia requiring medical management
* Individuals with severe chronic diseases, extensive extra-cardiac syndromes, or history of any cancer
* Individuals with current IV inotrope requirements
* Individuals with bleeding disorders or history of thrombosis
* Subjects not eligible for MRI or CT examination due to either a medical contraindication, including acute or chronic renal failure
* Individuals with a currently active infection being treated with oral antibiotics
* Individuals with the following conditions within 60 days prior to Ebstein repair surgery:

  * Cardiogenic shock or extracorporeal circulation
  * Documented infection requiring treatment with intravenous antibiotics
  * Cardiac condition requiring emergency procedure
  * Current or uncontrolled seizures or neurological injury that has resulted in a persistent deficit
  * Multi-system organ failure including acute or chronic renal failure
* Female subjects 10 years and older with positive pregnancy test or lack of effective birth control method during the 30 days prior to surgical Ebstein repair
* Individuals who weigh more than 90 kg

Ages: 6 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2016-09; Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Number of adverse events from time of index procedure | 24 months post index procedure
  Safety assessment of adverse events from time of index procedure will be analyzed by counts and percents using the chi-square test and Cochran-Armitage test for trends, and the two groups compared using the Fisher exact test. A Fisher's exact test with a 0.05 two-sided significance level will have 80% power to detect a difference in a sample size of 10 in each group. Thus having reasonable power to distinguish common rates for adverse events from very rare rates. Analysis of cardiac adverse events is in terms of the yes/no information at 24 months. Subjects will be censored upon lost to follow up. If some subjects are lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method and comparison between the two groups using the log-rank test. A confidence interval for the difference between groups will be given.
Severity of adverse events from time of index procedure | 24 months post index procedure
  Safety assessment of severity of adverse events from time of index procedure will be analyzed by counts and percents using the chi-square test and Cochran-Armitage test for trends, and the two groups compared using the Fisher exact test. A Fisher's exact test with a 0.05 two-sided significance level will have 80% power to detect a difference in a sample size of 10 in each group. Thus having reasonable power to distinguish common rates for adverse events from very rare rates. Subjects will be censored upon lost to follow up. If some subjects are lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method and comparison between the two groups using the log-rank test. A confidence interval for the difference between groups will be given.
Number of subjects who died | 24 months post index procedure
  Safety assessment of all-cause mortality will be analyzed by counts and percents using the chi-square test and Cochran-Armitage test for trends, and the two groups compared using the Fisher exact test. A Fisher's exact test with a 0.05 two-sided significance level will have 80% power to detect a difference in a sample size of 10 in each group. Thus having reasonable power to distinguish common rates for adverse events from very rare rates. Subjects will be censored upon lost to follow up. If some subjects are lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method and comparison between the two groups using the log-rank test. A confidence interval for the difference between groups will be given.
Number of subjects with sustained symptomatic cardiac arrhythmias | 24 months post index procedure
  Safety assessment of sustained symptomatic cardiac arrhythmias will be analyzed by counts and percents using the chi-square test and Cochran-Armitage test for trends, and the two groups compared using the Fisher exact test. A Fisher's exact test with a 0.05 two-sided significance level will have 80% power to detect a difference in a sample size of 10 in each group. Thus having reasonable power to distinguish common rates for adverse events from very rare rates. Subjects will be censored upon lost to follow up. If some subjects are lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method and comparison between the two groups using the log-rank test. A confidence interval for the difference between groups will be given.
Number of subjects with myocardial infarction | 24 months post index procedure
  Safety assessment of myocardial infarctions will be analyzed by counts and percents using the chi-square test and Cochran-Armitage test for trends, and the two groups compared using the Fisher exact test. A Fisher's exact test with a 0.05 two-sided significance level will have 80% power to detect a difference in a sample size of 10 in each group. Thus having reasonable power to distinguish common rates for adverse events from very rare rates. Subjects will be censored upon lost to follow up. If some subjects are lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method and comparison between the two groups using the log-rank test. A confidence interval for the difference between groups will be given.
Number of subjects with unexpected, invasive cardiovascular procedures | 24 months post index procedure
  Safety assessment of unexpected, invasive cardiovascular procedures will be analyzed by counts and percents using the chi-square test and Cochran-Armitage test for trends, and the two groups compared using the Fisher exact test. A Fisher's exact test with a 0.05 two-sided significance level will have 80% power to detect a difference in a sample size of 10 in each group. Thus having reasonable power to distinguish common rates for adverse events from very rare rates. Subjects will be censored upon lost to follow up. If some subjects are lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method and comparison between the two groups using the log-rank test. A confidence interval for the difference between groups will be given.
Number of serious adverse events | 24 months post index procedure
  Safety assessment of serious adverse events will be analyzed by counts and percents using the chi-square test and Cochran-Armitage test for trends, and the two groups compared using the Fisher exact test. A Fisher's exact test with a 0.05 two-sided significance level will have 80% power to detect a difference in a sample size of 10 in each group. Thus having reasonable power to distinguish common rates for adverse events from very rare rates. Subjects will be censored upon lost to follow up. If some subjects are lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method and comparison between the two groups using the log-rank test. A confidence interval for the difference between groups will be given.
Percentage of subjects in the treatment group that have cells delivered | 24 months post index procedure
  Feasibility of the BM-MNC cell therapy will be evaluated comparing number of subjects enrolled in the treatment group to subjects in the treatment group who are accrued and have cells delivered by percentage using the binomial distribution and exact confidence limits given.
Percentage of subjects in the treatment group completing the 24 month follow-up | 24 months post index procedure
  Feasibility of the BM-MNC cell therapy will be evaluated comparing number of subjects enrolled in the treatment group to subjects in the treatment group who are accrued and have cells delivered, who complete the 24 month follow-up visit by percentage.
Incidence of cardiac related hospitalizations from time of Ebstein repair | 1, 6, and 24 months post index procedure
  Efficacy will be evaluated using analysis of covariance (ANCOVA) from baseline to 24 months post-index procedure comparing outcomes between the treatment group to the control group. A sample size of 10 in each group using t-test will have 80% power to detect an effect size of 1.325 with a 0.050 two-sided significance level to identify a difference between means from the two groups. Descriptive statistics such as mean, median, SD, min, max, and 95% confidence intervals of the mean, and frequency distributions will be calculated for all variables by group. Fisher exact test will have 80% power to detect a difference in a sample size of 10 in each group having reasonable power to distinguish common rates from very rare rates. Analysis is in terms of the yes/no information at 24 months. Subjects will be censored upon lost to follow up. If a subject is lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method.
Incidence of cardiac arrhythmias from time of index procedure | 1, 6, and 24 months post index procedure
  Efficacy will be evaluated using analysis of covariance (ANCOVA) from baseline to 24 months post-index procedure comparing outcomes between the treatment group to the control group. A sample size of 10 in each group using t-test will have 80% power to detect an effect size of 1.325 with a 0.050 two-sided significance level to identify a difference between means from the two groups. Descriptive statistics such as mean, median, SD, min, max, and 95% confidence intervals of the mean, and frequency distributions will be calculated for all variables by group. Fisher exact test will have 80% power to detect a difference in a sample size of 10 in each group having reasonable power to distinguish common rates from very rare rates. Analysis is in terms of the yes/no information at 24 months. Subjects will be censored upon lost to follow up. If a subject is lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method.
Change in CT derived right ventricular dimensions from time of pre-operative evaluation | 6 and 24 months post index procedure
  Efficacy will be evaluated using analysis of covariance (ANCOVA) from baseline to 24 months post-index procedure comparing outcomes between the treatment group to the control group. End volume measurements recorded using mL and indexed to body surface area (BSA) using mL/m^2.A sample size of 10 in each group using t-test will have 80% power to detect an effect size of 1.325 with a 0.050 two-sided significance level to identify a difference between means from the two groups. Descriptive statistics such as mean, median, SD, min, max, and 95% confidence intervals of the mean, and frequency distributions will be calculated for all variables by group. Fisher exact test will be used to distinguish common rates from very rare rates. Analysis is in terms of yes/no information at 24 months.If a subject is lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method.
Change in echocardiography derived cardiac output from time of pre-operative evaluation | 1, 6, and 24 months post index procedure
  Efficacy will be evaluated using analysis of covariance (ANCOVA) from baseline to 24 months post-index procedure comparing outcomes between the treatment group to the control group.Volume is measured in L/min and Volume Index is L/min/m^2.Using t-test will have 80% power to identify a difference between means from the two groups. Descriptive statistics such as mean, median, SD, min, max, and 95% confidence intervals of the mean, and frequency distributions will be calculated for all variables by group. Fisher exact test will have 80% power to detect a difference in a sample size of 10 in each group to distinguish common rates from very rare rates. Analysis in terms of yes/no information at 24 months. If a subject is lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method.
Change in NT-Pro-BNP derived cardiac function trend from time of pre-operative evaluation | During hospitalization up to 29 days, 1, 6 and 24 months post index procedure
  Efficacy will be evaluated using analysis of covariance (ANCOVA) from baseline to 24 months post-index procedure comparing outcomes between the treatment group to the control group. A sample size of 10 in each group using t-test will have 80% power to detect an effect size of 1.325 with a 0.050 two-sided significance level to identify a difference between means from the two groups. Descriptive statistics such as mean, median, SD, min, max, and 95% confidence intervals of the mean, and frequency distributions will be calculated for all variables by group. Fisher exact test will have 80% power to detect a difference in a sample size of 10 in each group having reasonable power to distinguish common rates from very rare rates. Analysis is in terms of the yes/no information at 24 months. Subjects will be censored upon lost to follow up. If a subject is lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method.
Incidence of cardiac related hospitalizations in the treatment group from time of pre-operative evaluation compared to the control group | 1, 6, and 24 months post index procedure
  Efficacy will be evaluated using analysis of covariance (ANCOVA) from baseline to 24 months post-index procedure comparing outcomes between the treatment group to the control group. A sample size of 10 in each group using t-test will have 80% power to detect an effect size of 1.325 with a 0.050 two-sided significance level to identify a difference between means from the two groups. Descriptive statistics such as mean, median, SD, min, max, and 95% confidence intervals of the mean, and frequency distributions will be calculated for all variables by group. Fisher exact test will have 80% power to detect a difference in a sample size of 10 in each group having reasonable power to distinguish common rates from very rare rates. Analysis is in terms of the yes/no information at 24 months. Subjects will be censored upon lost to follow up. If a subject is lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method.
Incidence of cardiac arrhythmias in the treatment group from time of pre-operative evaluation compared to the control group | 1, 6, and 24 months post index procedure
  Efficacy will be evaluated using analysis of covariance (ANCOVA) from baseline to 24 months post-index procedure comparing outcomes between the treatment group to the control group. A sample size of 10 in each group using t-test will have 80% power to detect an effect size of 1.325 with a 0.050 two-sided significance level to identify a difference between means from the two groups. Descriptive statistics such as mean, median, SD, min, max, and 95% confidence intervals of the mean, and frequency distributions will be calculated for all variables by group. Fisher exact test will have 80% power to detect a difference in a sample size of 10 in each group having reasonable power to distinguish common rates from very rare rates. Analysis is in terms of the yes/no information at 24 months. Subjects will be censored upon lost to follow up. If a subject is lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method.
Change in MRI derived cardiac output in the treatment group from time of pre-operative evaluation compared to the control group | 6 and 24 months post index procedure
  Efficacy will be evaluated using analysis of covariance (ANCOVA) from baseline to 24 months post-index procedure comparing outcomes between the treatment group to the control group.Volume is measured in L/min and Volume Index is L/min/m^2.Using t-test will have 80% power to identify a difference between means from the two groups. Descriptive statistics such as mean, median, SD, min, max, and 95% confidence intervals of the mean, and frequency distributions will be calculated for all variables by group. Fisher exact test will have 80% power to detect a difference in a sample size of 10 in each group to distinguish common rates from very rare rates. Analysis in terms of yes/no information at 24 months.If a subject is lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method.
Change in echocardiography derived right ventricular dimensions from time of pre-operative evaluation | 1, 6, and 24 months post index procedure
  Efficacy will be evaluated using analysis of covariance (ANCOVA) from baseline to 24 months post-index procedure comparing outcomes between the treatment group to the control group. End volume measurements recorded using mL and indexed to body surface area (BSA) using mL/m^2,diameter as cm.A sample size of 10 in each group using t-test will have 80% power to detect an effect size of 1.325 with a 0.050 two-sided significance level to identify a difference between means from the two groups. Descriptive statistics such as mean, median, SD, min, max, and 95% confidence intervals of the mean, and frequency distributions will be calculated for all variables by group. Fisher exact test will be used to distinguish common rates from very rare rates. Analysis is in terms of yes/no information at 24 months.If a subject is lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method.
Change in NT-Pro-BNP derived cardiac function trend in the treatment group from time of pre-operative evaluation compared to the control group | During hospitalization up to 29 days, 1, 6, and 24 month post index procedure
  Efficacy will be evaluated using analysis of covariance (ANCOVA) from baseline to 24 months post-index procedure comparing outcomes between the treatment group to the control group. A sample size of 10 in each group using t-test will have 80% power to detect an effect size of 1.325 with a 0.050 two-sided significance level to identify a difference between means from the two groups. Descriptive statistics such as mean, median, SD, min, max, and 95% confidence intervals of the mean, and frequency distributions will be calculated for all variables by group. Fisher exact test will have 80% power to detect a difference in a sample size of 10 in each group having reasonable power to distinguish common rates from very rare rates. Analysis is in terms of the yes/no information at 24 months. Subjects will be censored upon lost to follow up. If a subject is lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method.
Number of serious adverse events from time of enrollment | index procedure
  Safety assessment of the number of serious adverse events from time of enrollment will be analyzed by counts and percents using the chi-square test and Cochran-Armitage test for trends, and the two groups compared using the Fisher exact test. A Fisher's exact test with a 0.05 two-sided significance level will have 80% power to detect a difference in a sample size of 10 in each group. Thus having reasonable power to distinguish common rates for adverse events from very rare rates. Subjects will be censored upon lost to follow up. If some subjects are lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method and comparison between the two groups using the log-rank test. A confidence interval for the difference between groups will be given.
Percentage of subjects in the treatment group whose cells meet all release criteria | 24 months post index procedure
  Feasibility of the BM-MNC cell therapy will be evaluated comparing number of subjects enrolled in the treatment group to subjects in the treatment group with collected bone marrow and the bone marrow cells have met all product release criteria to any products that did not meet release criteria by percentage.
Change in CT derived cardiac output from time of pre-operative evaluation | 6 and 24 months post index procedure
  Efficacy will be evaluated using analysis of covariance (ANCOVA) from baseline to 24 months post-index procedure comparing outcomes between the treatment group to the control group.Volume is measured in L/min and Volume Index is L/min/m^2.Using t-test will have 80% power to identify a difference between means from the two groups. Descriptive statistics such as mean, median, SD, min, max, and 95% confidence intervals of the mean, and frequency distributions will be calculated for all variables by group. Fisher exact test will have 80% power to detect a difference in a sample size of 10 in each group to distinguish common rates from very rare rates. Analysis in terms of yes/no information at 24 months. If a subject is lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method.
Change in MRI derived right ventricle ejection fraction in the treatment group from time of pre-operative evaluation compared to the control group | 6 and 24 months post index procedure
  Efficacy will be evaluated using analysis of covariance (ANCOVA) from baseline to 24 months post-index procedure comparing outcomes between the treatment group to the control group measured in %.Using t-test will have 80% power to detect an effect size of 1.325 with a 0.050 two-sided significance level to identify a difference between means from the two groups. Descriptive statistics such as mean, median, SD, min, max, and 95% confidence intervals of the mean, and frequency distributions will be calculated for all variables by group. Fisher exact test will have 80% power to detect a difference in a sample size of 10 in each group having reasonable power to distinguish common rates from very rare rates. Analysis is in terms of the yes/no information at 24 months. Subjects will be censored upon lost to follow up. If a subject is lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method.
Change in MRI derived right ventricular dimensions in the treatment group from time of pre-operative evaluation compared to the control group | 6 and 24 months post index procedure
  Efficacy will be evaluated using analysis of covariance (ANCOVA) from baseline to 24 months post-index procedure comparing outcomes between the treatment group to the control group. End volume measurements recorded using mL and indexed to body surface area (BSA) using mL/m^2.A sample size of 10 in each group using t-test will have 80% power to detect an effect size of 1.325 with a 0.050 two-sided significance level to identify a difference between means from the two groups. Descriptive statistics such as mean, median, SD, min, max, and 95% confidence intervals of the mean, and frequency distributions will be calculated for all variables by group. Fisher exact test will be used to distinguish common rates from very rare rates. Analysis is in terms of yes/no information at 24 months.If a subject is lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method.
Change in CT derived right ventricle ejection fraction from time of pre-operative evaluation | 6 and 24 months post index procedure
  Efficacy will be evaluated using analysis of covariance (ANCOVA) from baseline to 24 months post-index procedure comparing outcomes between the treatment group to the control group measured in %.Using t-test will have 80% power to detect an effect size of 1.325 with a 0.050 two-sided significance level to identify a difference between means from the two groups. Descriptive statistics such as mean, median, SD, min, max, and 95% confidence intervals of the mean, and frequency distributions will be calculated for all variables by group. Fisher exact test will have 80% power to detect a difference in a sample size of 10 in each group having reasonable power to distinguish common rates from very rare rates. Analysis is in terms of the yes/no information at 24 months. Subjects will be censored upon lost to follow up. If a subject is lost to follow-up then fractions at 24 months will be described using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Y Qureshi, MBBS, Principal Investigator — Mayo Clinic; Timothy J Nelson, MD, PhD, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Leary PW, Qureshi MY, Cetta F, Nelson TJ, Holst KA, Dearani JA; Wanek Program Clinical Pipeline Group. Cone Reconstruction for Ebstein Anomaly: Ventricular Remodeling and Preliminary Impact of Stem Cell Therapy. Mayo Clin Proc. 2021 Dec;96(12):3053-3061. doi: 10.1016/j.mayocp.2021.02.015. Epub 2021 Sep 1. PMID 34479739
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials